CLINICAL TRIAL: NCT00005719
Title: Sustaining Women's Smoking Cessation Postpartum
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4928; R01HL044898 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Lung Diseases; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Lung Diseases; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To conduct a five-year demonstration and education project to sustain smoking cessation postpartum by women who had stopped smoking in pregnancy.

DETAILED DESCRIPTION:
BACKGROUND:

The results from this study were expected to demonstrate the effectiveness of a practical program to protect women and their families from direct and indirect smoke exposure and to contribute longitudinal data on change processes involved in smoking cessation, especially those over the maintenance, relapse, and recycling stages, in a relatively complete population through a critical transition.

DESIGN NARRATIVE:

The TLC Program, unique in its focus on the postpartum period, used a researched model of behavior change that matched messages and skill training with the woman's stage of change. It also addressed the whole family to create a supportive environment for individual change, included other steps for families to protect children from passive smoke and negative modeling, and focused on smoking and smoke exposure directly as well as through self-care and child-care messages. The program used innovative materials, including videotapes and intervention.

The study took place in two multi-ethnic health-care sites where the research team had conducted previous studies. The study used a randomized mixed design with 500 women who smoked regularly before pregnancy and who had been abstinent for > 30 days at their 28th week of pregnancy. The primary outcome was abstinence at one year postpartum. Secondary outcomes were partner smoking status and exposure of the index baby. Self report was validated biochemically in samples of mothers and babies. The study design separated data collection from the experiments by enrolling subjects in a university-sponsored study of new mothers' health-care site.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 1996-06

REFERENCES:
- [Background] Dolan-Mullen P, Ramirez G, Groff JY. A meta-analysis of randomized trials of prenatal smoking cessation interventions. Am J Obstet Gynecol. 1994 Nov;171(5):1328-34. doi: 10.1016/0002-9378(94)90156-2. PMID 7977542
- [Background] Mullen PD, Simons-Morton DG, Ramirez G, Frankowski RF, Green LW, Mains DA. A meta-analysis of trials evaluating patient education and counseling for three groups of preventive health behaviors. Patient Educ Couns. 1997 Nov;32(3):157-73. doi: 10.1016/s0738-3991(97)00037-2. PMID 9423498
- [Background] Groff JY, Mullen PD, Mongoven M, Burau K. Prenatal weight gain patterns and infant birthweight associated with maternal smoking. Birth. 1997 Dec;24(4):234-9. doi: 10.1111/j.1523-536x.1997.tb00596.x. PMID 9460314
- [Background] Hudmon KS, Mullen PD, Nicol L, Hammond SK, Sockrider MM, Sajak T, Thompson J. Telephone-guided placement and removal of nicotine monitors for the assessment of passive exposure to environmental tobacco smoke. Toxicol Ind Health. 1997 Jan-Feb;13(1):73-80. doi: 10.1177/074823379701300107. PMID 9098952
- [Background] Stotts AL, DiClemente CC, Carbonari JP, Mullen PD. Pregnancy smoking cessation: a case of mistaken identity. Addict Behav. 1996 Jul-Aug;21(4):459-71. doi: 10.1016/0306-4603(95)00082-8. PMID 8830904
- [Background] Stotts AL, DiClemente CC, Carbonari JP, Mullen PD. Postpartum return to smoking: staging a "suspended" behavior. Health Psychol. 2000 Jul;19(4):324-32. doi: 10.1037//0278-6133.19.4.324. PMID 10907650